CLINICAL TRIAL: NCT03453710
Title: Arthroscopic Bankart Repair and Remplissage Versus Latarjet Coracoid Transfer for Recurrent Anterior Glenohumeral Instability With Subcritical Bone Loss - A Randomized Controlled Trial
Brief Title: Remplissage Versus Latarjet Coracoid Transfer for Recurrent Shoulder Instability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Panam Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111328
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Shoulder Dislocation
Keywords: Bankart Repair; Remplissage; Latarjet coracoid transfer
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Patients will be evaluated by a blinded study nurse, unaware of treatment allocation, for administration of baseline questionnaires, as well as subsequent post-operative questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bankart Repair and Remplissage (Active Comparator): Patients randomized to the all-arthroscopic group (Bankart repair and remplissage) will undergo a standard arthroscopic anterior labral repair with a minimum of 3 suture anchors, followed by remplissage with 1 or 2 anchors, at the discretion of the treating surgeon.
  Interventions: Procedure: Bankart Repair plus Remplissage
- Latarjet Coracoid Transfer (Active Comparator): Patients randomized to the open Latarjet coracoid transfer will undergo a Latarjet coracoid transfer through a deltopectoral approach and horizontal split in the subscapularis at the superior 2/3, inferior 1/3 junction. The coracoid process will be oriented in the conventional manner, with the inferior surface against the glenoid vault, secured with two cannulated screws
  Interventions: Procedure: Latarjet coracoid transfer

INTERVENTIONS:
Procedure: Bankart Repair plus Remplissage — Arthroscopic Bankart repair with a minimum of 3 anchors
  1 or 2 anchor Remplissage subsequently performed with percutaneous anchor insertion in the base of the Hill-Sachs defect, and sutures passed in a horizontal mattress configuration 1 cm apart, tied in the subacromial space.
  Arms: Bankart Repair and Remplissage
Procedure: Latarjet coracoid transfer — Coracoid transfer performed via deltopectoral approach with horizontal subscapularis split. Graft placed in the conventional orientation, secured with 2 screws, ensuring the graft is not lateral to the glenoid rim.
  Arms: Latarjet Coracoid Transfer

SUMMARY:
This is a pilot study designed as a prospective, randomized controlled trial comparing arthroscopic Bankart repair and Remplissage with an open Latarjet coracoid transfer for the treatment of recurrent anterior glenohumeral instability with subcritical bone loss.

DETAILED DESCRIPTION:
Presently, consensus guidelines for the surgical management of anterior glenohumeral instability are lacking. While there has been continual evolution in available arthroscopic instrumentation, this has not translated to improvements in patient outcomes. Isolated arthroscopic bankart repair is often associated with unacceptably high rates of failure, with a recent systematic review identifying continued recurrence rates of 14.2%. Improved recognition of bone defects and identification of critical defect sizes that contribute to recurrent instability and failed stabilization have lead to improvements in treatment algorithms. It has been widely accepted that glenoid defects exceeding 20% of anteroposterior (AP) width and humeral head defects exceeding 30% of the humeral head width contribute to recurrent instability. For defects of this magnitude, isolated arthroscopic Bankart repair is insufficient in restoring joint stability, and more extensive procedures are required. This can include adding a remplissage to the arthroscopic Bankart repair or open allograft reconstruction for humeral defects; or Latarjet coracoid transfer for glenoid defects.

However, often patients present with combined 'bipolar' bone loss, where individual defects are subcritical in size. There is increasing recognition that the presence of this combined bone loss may lead to increased rates of failure with an isolated arthroscopic bankart repair. Currently, accepted treatment options for bipolar bone loss include a combined arthroscopic Bankart repair and remplissage, or a Latarjet coracoid transfer. While there is supportive biomechanical data for each procedure, and limited case series in the literature, there remains a paucity of high-quality evidence to guide treatment for this complex clinical scenario. Consequently, we aim to perform a pilot study designed as a prospective, randomized controlled trial comparing arthroscopic Bankart repair and Remplissage with an open Latarjet coracoid transfer.

ELIGIBILITY:
Inclusion Criteria:

* anterior shoulder instability (>1 dislocation)
* age >14 years
* evidence of a Hill-Sachs defect on MRI or CT,
* < 20% anteroposterior glenoid bone loss

Exclusion Criteria:

* >20% anteroposterior glenoid bone loss
* significant shoulder comorbidities (i.e., osteoarthritis, previous surgery other than previous instability), active joint or systemic infection, significant muscle paralysis, rotator cuff or Charcot's arthropathy,
* significant medical comorbidity that may alter effectiveness of surgical intervention
* major medical illness,
* unable to speak French or English,
* psychiatric illness that precludes informed consent,
* unwilling to be followed for 2 years

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Western Ontario Shoulder Instability (WOSI) Score | 24 months
  Western Ontario Shoulder Instability (WOSI) questionnaire is a tool designed for self-assessment of shoulder function for patients with instability problems. Difference between study arm outcomes will be assessed using pre-op and post-op WOSI score as a covariate.
  This questionnaire has 21 questions, each scored on a scale from 0 to 100, with 0 being the best score (no limitations related to the shoulder) and 100 representing the worst score.
  Overall, the questionnaire is scored as a percentage of the maximum score of 2100 points.
  There are subscale components reporting on: physical symptoms (questions 1 through 10; maximum score of 1000); sports/recreation/work (questions 11 through 14; maximum score 400); lifestyle (questions 15 through 18; maximum score 400); and emotion (questions 19-21; maximum score 300).
  Subscale scores are added to determine the total score out of a possible 2100 points, with 2100, or 100%, representing the worst possible score.

SECONDARY OUTCOMES:
Pain numeric rating scale (NRS) | 24 months
  This tool is designed to evaluate pain. The Scale is from 0-100 to determine shoulder pain pre and post-operatively; 0=extreme pain, 100=no pain
Simple Shoulder Test (SST) | 24 months
  Simple Shoulder Test (SST) is a series of 12 "yes" or "no" questions the patient answers about the function of the involved shoulder. The answers to these questions provides a standardized way of recording the function of a shoulder before and after treatment. Differences between study arm outcomes will be assessed using pre-op SST scores as a covariate
American Shoulder and Elbow Society (ASES) assessment | 24 months
  The ASES assessment (patient report section) is a region-specific questionnaire designed for self-assessment of aspects of pain and function. Difference between study arm outcomes will be assessed using pre-op ASES score as a covariate
Range of motion | 24 months
  Range of motion will be evaluated using a goniometer to calculate: forward flexion, abduction, external rotation and internal rotation
Post-operative complications | 24 months
  Post-surgical complications will be collected including: neurologic injury (neuropraxia); superficial wound infection; deep surgical site infection; coracoid non-union or malunion; posterior shoulder pain; stiffness; recurrent instability

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Pan Am Clinic, Winnipeg, Manitoba
  - Fowler Kennedy Sport Medicine Clinic, London, Ontario

IPD SHARING:
Plan to Share IPD: No